CLINICAL TRIAL: NCT04909463
Title: Effects of Using the Duracore Splinting Device on Patient Outcomes Related to Chest Trauma
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Limited resources
Sponsor: CommonSpirit Health (Other)
Responsible Party: Principal Investigator, Trenton Bradbury, Registered Respiratory Therapist, CommonSpirit Health
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 1517921
Record Dates: First submitted 2021-01-04; First posted 2021-06-01 (Actual); Results first posted 2025-05-14 (Actual); Last update posted 2025-05-14 (Actual); Status verified 2025-04

CONDITIONS: Rib Fractures; Rib Fracture Multiple
MeSH Terms: conditions — Rib Fractures

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (4):
- Unilateral rib fractures only, no device intervention (No Intervention): Unilateral rib fractures only, no device intervention
- Unilateral rib fractures, device intervention (Experimental): Unilateral rib fractures, will receive device intervention
  Interventions: Device: Chest Splint
- Bilateral rib fractures, no device intervention (No Intervention): Bilateral rib fractures, no device intervention
- Bilateral rib fractures, device intervention (Experimental): Bilateral rib fractures, will receive device intervention
  Interventions: Device: Chest Splint

INTERVENTIONS:
Device: Chest Splint — Those receiving intervention will be given the Duracore chest splint for use throughout the trial.
  Other Names: Duracore
  Arms: Bilateral rib fractures, device intervention; Unilateral rib fractures, device intervention

SUMMARY:
The purpose of this study is to use the Duracore splinting device to measure lung capacities of patients with rib fractures in control and experimental groups to determine if lung capacities improve with the splint.

DETAILED DESCRIPTION:
The purpose of this study is to use the Duracore patient operated torso splinting device for patients with chest trauma, including rib fractures, to improve deep breathing and help with reduced hospital length of stays (LOS). The hypothesis of this study is that the use of the Duracore splinting device will reduce hospital length of stays and improve patient lung capacities over the course of admission following chest trauma.

The study will use a randomized-experimental design and will be randomized via envelope randomization, with experimenters being blinded. A total of 104 patients, 26 in each group, will undergo initial incentive spirometry and forced vital capacity (FVC) and forced expiratory volume at 1 second (FEV1) tests. Number of subjects to be used are 150 to account for withdrawals, incomplete data sets, extraneous results, etc. Groups will consist of a control versus experimental group, stratified into bilateral and unilateral rib fractures. Three days' worth of data will be collected for each of the tests and will also be collected 24 hours prior to discharge. Length of stays will be compared for experimental and control groups, as well as time to ambulation (collected from the first physical therapy assessment). Injury severity score will also be collected to determine any correlation by severity of injury. Patient satisfaction surveys for the device will also be collected to determine if the patients feel a difference with the device.

Little research as been conducted to determine the significance of a splinting device used in patients with chest trauma, and it is still uncertain whether these devices improve overall patient outcomes. Contradicting studies with similar experimental designs show either some significance (p-value) or insignificance in pulmonary function pre- and post-treatment. This gap in current knowledge leaves room for concern in whether the patient truly benefits from a splinting device in this type of injury. Changes in FVC/FEV1 ratio in this patient population are not readily demonstrated in most of these studies, as well as differing length of stays. This study will contribute to this base of knowledge by determining the effects of the Duracore splinting device on this patient population using the objectives.

ELIGIBILITY:
Inclusion:

* Adult patient admitted to the trauma service at Penrose Hospital
* Willing and able to comply with all requirements of the study
* Active diagnosis of rib fractures
* Male or female 18 years and older
* Able to provide written informed consent to participate in the study
* Must be physically able to don and use the splinting device independently without assistance.

Exclusion:

* <18 years old
* History of pulmonary disease, lobectomy, or lung transplant
* Current smoker of tobacco products
* Diagnosis of flail chest
* Pregnant Women
* Prisoners
* Cognitively Impaired; must be alert and oriented x 3

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2020-12-04 (Actual); Primary Completion 2021-07-30 (Actual); Study Completion 2021-07-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Trenton Bradbury, BS, Principal Investigator — CommonSpirit Health
Locations (1):
- Penrose Hospital, Colorado Springs, Colorado, United States

IPD SHARING:
Plan to Share IPD: No
No IPD will be shared. All information pertaining to statistical significance or lack thereof will be outlined in the final study publication.

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Unilateral Rib Fractures Only, no Device Intervention | Unilateral Rib Fractures, Device Intervention | Bilateral Rib Fractures, no Device Intervention | Bilateral Rib Fractures, Device Intervention
Started | 3 | 4 | 1 | 0
Completed | 1 | 2 | 0 | 0
Not Completed | 2 | 2 | 1 | 0
Not completed — Withdrawal by Subject | 0 | 1 | 0 | 0
Not completed — Lost to Follow-up | 2 | 1 | 1 | 0

BASELINE CHARACTERISTICS:
Population: lack of available subjects due to the covid19 pandemic
Groups:
- Total: Total of all reporting groups
Arm/Group | Unilateral Rib Fractures Only, no Device Intervention | Unilateral Rib Fractures, Device Intervention | Bilateral Rib Fractures, no Device Intervention | Bilateral Rib Fractures, Device Intervention | Total
Number analyzed (Participants) | 3 | 4 | 1 | 0 | 8
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 1 | 3 | 1 |  | 5
  >=65 years | 2 | 1 | 0 |  | 3
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 2 | 0 |  | 4
  Male | 1 | 2 | 1 |  | 4
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: FVC Change
Description: Change in forced vital capacities over time using the device as compared to control groups
Time Frame: 3 days of consistent measuring and a final measurement 24 hours prior to expected discharge
Population: Eight participants were enrolled before early termination of the study due to the COVID-19 pandemic. Three participants contributed data for this outcome measure. Two participants were assigned to the Unilateral Rib Fractures with Device Intervention group and one participant to the Unilateral Rib Fractures without Device group. Five participants withdrew early or were discharged without providing complete outcome data. Results are summarized only for participants who contributed data.
Measure: Mean (Standard Deviation); unit: Liters (L)
Arm/Group | Unilateral Rib Fractures Only, no Device Intervention | Unilateral Rib Fractures, Device Intervention | Bilateral Rib Fractures, no Device Intervention | Bilateral Rib Fractures, Device Intervention
Number analyzed (Participants) | 1 | 2 | 0 | 0
Liters (L) | 0.06 (0) | 0.34 (0.33) |  |

2. Primary Outcome: FEV1 Change
Description: Change in forced expiratory volume in one second over hospital duration using the device as compared to control groups
Time Frame: 3 days of consistent measuring and a final measurement 24 hours prior to expected discharge
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Liters (L)
Arm/Group | Unilateral Rib Fractures Only, no Device Intervention | Unilateral Rib Fractures, Device Intervention | Bilateral Rib Fractures, no Device Intervention | Bilateral Rib Fractures, Device Intervention
Number analyzed (Participants) | 1 | 2 | 0 | 0
Liters (L) | 0.03 (0) | 0.33 (0.46) |  |

3. Primary Outcome: FEV1 Percent Change
Description: Change in FEV1/FVC ratio (expressed as FEV1%) over hospital duration using the device as compared to control groups
Time Frame: 3 days of consistent measuring and a final measurement 24 hours prior to expected discharge
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Percentage (%)
Arm/Group | Unilateral Rib Fractures Only, no Device Intervention | Unilateral Rib Fractures, Device Intervention | Bilateral Rib Fractures, no Device Intervention | Bilateral Rib Fractures, Device Intervention
Number analyzed (Participants) | 1 | 2 | 0 | 0
Percentage (%) | -0.63 (0) | 4.49 (12.40) |  |

4. Secondary Outcome: Length of Stay
Description: The length of stay for the entire admission to the time of discharge
Time Frame: Documented at time of discharge, assessed up to 14 days.
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | Unilateral Rib Fractures Only, no Device Intervention | Unilateral Rib Fractures, Device Intervention | Bilateral Rib Fractures, no Device Intervention | Bilateral Rib Fractures, Device Intervention
Number analyzed (Participants) | 1 | 2 | 0 | 0
Days | 2 (0) | 4.5 (2.12) |  |

5. Secondary Outcome: Time to Ambulation
Description: The initial time of ambulation documented after admission.
Time Frame: 0-48 hours after admission.
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Hours
Arm/Group | Unilateral Rib Fractures Only, no Device Intervention | Unilateral Rib Fractures, Device Intervention | Bilateral Rib Fractures, no Device Intervention | Bilateral Rib Fractures, Device Intervention
Number analyzed (Participants) | 1 | 2 | 0 | 0
Hours | 19.8 (0) | 22.75 (3.46) |  |

6. Secondary Outcome: Injury Severity Score
Description: Use of the Injury Severity Score to measure the degree of injury and how it affects outcomes associated with the chest splint. This is measured on a scale from 1 to 6; 1 being relatively minor and 6 being untreatable.
Time Frame: Documented within 2 weeks of admission date.
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score
Arm/Group | Unilateral Rib Fractures Only, no Device Intervention | Unilateral Rib Fractures, Device Intervention | Bilateral Rib Fractures, no Device Intervention | Bilateral Rib Fractures, Device Intervention
Number analyzed (Participants) | 1 | 2 | 0 | 0
score | 9 (0) | 2.5 (2.12) |  |

7. Secondary Outcome: Day of Admission
Description: Documenting date and time of admission
Time Frame: Within first 24 hours of admission
Population: Eight participants were enrolled before early termination of the study due to the COVID-19 pandemic. Three participants contributed admission date and time documentation for this outcome measure. Two participants were assigned to the Unilateral Rib Fractures with Device Intervention group and one participant to the Unilateral Rib Fractures without Device group. Date and time of admission were recorded for clinical documentation purposes. No statistical analysis was performed for this outcome.
Measure: Count of Participants; unit: Participants
Arm/Group | Unilateral Rib Fractures Only, no Device Intervention | Unilateral Rib Fractures, Device Intervention | Bilateral Rib Fractures, no Device Intervention | Bilateral Rib Fractures, Device Intervention
Number analyzed (Participants) | 1 | 2 | 0 | 0
Participants | 1 | 2 |  |

8. Secondary Outcome: Vital Capacity Measurement Via Incentive Spirometry
Description: Change in vital capacity values indicating changes in deep breathing over the course of hospitalization while using the Duracore device
Time Frame: 3 days of consistent measuring and a final measurement 24 hours prior to expected discharge
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Liters (L)
Arm/Group | Unilateral Rib Fractures Only, no Device Intervention | Unilateral Rib Fractures, Device Intervention | Bilateral Rib Fractures, no Device Intervention | Bilateral Rib Fractures, Device Intervention
Number analyzed (Participants) | 1 | 2 | 0 | 0
Liters (L) | 0.20 (0) | 0.95 (0.21) |  |

ADVERSE EVENTS:
Time Frame: 7 months
Description: The number of participants at risk for serious adverse events, all-cause mortality, and Other (Not Including Serious) Adverse Events is zero for Bilateral Rib Fractures, Device Intervention because there were no subjects in that arm.
Arm/Group | Unilateral Rib Fractures Only, no Device Intervention | Unilateral Rib Fractures, Device Intervention | Bilateral Rib Fractures, no Device Intervention | Bilateral Rib Fractures, Device Intervention
All-Cause Mortality (participants affected / at risk) | 0/3 | 0/4 | 0/1 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/3 | 0/4 | 0/1 | 0/0
Other Adverse Events (participants affected / at risk) | 0/3 | 0/4 | 0/1 | 0/0

LIMITATIONS AND CAVEATS:
Early termination due to subject unavailability due to the COVID-19 pandemic. Uninterpretable data.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-12-08): https://cdn.clinicaltrials.gov/large-docs/63/NCT04909463/Prot_SAP_000.pdf